CLINICAL TRIAL: NCT07002723
Title: Effects of Esketamine Combined With Dexmedetomidine on Postoperative Sleep Quality in Elderly Patients Undergoing Hip Surgery:A Superiority Randomized Controlled Trail
Brief Title: Effects of Esketamine Combined With Dexmedetomidine on Postoperative Sleep Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-045
Record Dates: First submitted 2025-05-11; First posted 2025-06-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-04

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine combined with dexmedetomidine group (Experimental): After successful neuraxial anesthesia, 0.125mg/kg esketamine and 0.3ug/kg dexmedetomidine were diluted into 30ml of normal saline and continuously pumped for 20 minutes, followed by a micropump: 15ug/kg/h esketamine 0.02ug/kg/h dexmedetomidine to 96ml saline, continuous amount: 2ml/h, continuous pumping for 48h.
  Interventions: Drug: Esketamine combined with dexmedetomidine
- Normal saline group (Placebo Comparator): After successful neuraxial anesthesia, 30ml of normal saline was continuously pumped for 20 minutes, followed by a micropump: 96ml of saline, continuous amount: 2ml/h for 48h.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Esketamine combined with dexmedetomidine — After successful neuraxial anesthesia, 0.125mg/kg esketamine and 0.3ug/kg dexmedetomidine are diluted into 30ml of normal saline and continuously pumped for 20 minutes, then connected to a micropump: 15ug/kg/h esketamine 0.02ug/kg/h dexmedetomidine to 96ml saline, continuous amount: 2ml/h, continuous pumping for 48h.
  Arms: Esketamine combined with dexmedetomidine group
Drug: Normal saline — After successful neuraxial anesthesia, 30ml of normal saline was continuously pumped for 20 minutes, followed by a micropump: 96ml of saline, continuous amount: 2ml/h for 48h.
  Arms: Normal saline group

SUMMARY:
1. Eligible patients are randomly divided into experimental and control groups；
2. The experimental group is given esketamine combined with dexmedetomidine，while the control group is given normal saline；
3. The patients' sleep, pain, and cognition are followed up after surgery.

DETAILED DESCRIPTION:
One day before surgery, the investigators collect baseline data from patients at the bedside. Preoperative sleep quality is assessed using Pittsburgh sleep quality index(PSQI); Three-Minute Confusion Assessment Method(3D-CAM)is used to assess the incidence of delirium; cognitive function is assessed using Montreal Cognitive Assessment(MoCA); The Hospital Anxiety and Depression Scale (HADS) is used to assess patients' mood; Wong-Baker faces pain scale revision(FPS-R) and Numeric Rating Scale(NRS) are used to assess the patient's pain score at rest and during activity, and laboratory tests (Hb, Alb, K, NA, Cr, Alb, e-GFR) are recorded.

On the day of surgery, after successful neuraxial anesthesia, in the experimental group ，0.125mg/kg esketamine and 0.3ug/kg dexmedetomidine are diluted into 30ml of normal saline and continuously pumped for 20 minutes, followed by a micropump: 15ug/kg/h esketamine 0.02ug/kg/h dexmedetomidine to 96ml saline, continuous amount: 2ml/h, continuous pumping for 48h. Morphine 1 mg is given epidural at the beginning of surgery；while in the control group, same amount of normal saline is given. The patients are followed up for sleep quality, pain and delirium incidence after surgery. Long-term telephone follow-up of patients are focused on their cognitive function and recovery quality.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 65 years old;
* Hip fracture surgery under neuraxial anesthesia;
* Signed informed consent.

Exclusion Criteria:

* ASA classification≥ Class V;
* Presence of neuraxial anesthesia contraindications: coagulation dysfunction, thrombocytopenia, neuraxial mass, puncture site infection, etc.;
* Patients with contraindications to esketamine (such as allergies, intracranial aneurysms, hyperthyroidism and glaucoma);
* Patients with contraindications to dexmedetomidine (allergies);
* Patients with severe cardiovascular diseases such as sick sinus syndrome, severe sinus bradycardia (heart rate < 50 beats/min), atrioventricular block grade II or above without pacemaker, unstable angina, severe valvular heart disease, severe arrhythmia, severe macrovascular disease with New York Heart Association class III patients, etc.;
* Obstructive sleep apnea syndrome (STOP-BANG score > 3 points);
* Patients with severe hepatic and renal insufficiency (such as Child-Pugh score III, creatinine clearance < 35 mL/min, preoperative dialysis);
* Those who have delirium, dementia, moderate to severe cognitive dysfunction and psychiatric disorders before the start of the trial and are unable to communicate and cooperate with the investigator.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
sleep quality | the first postoperative night
  Richards-Campbell sleep questionnaire (RCSQ) score is used to assess the sleep quality, the total score is 100 point, the lowest score is 0 point, and the highest score is 100 point, with higher scores representing better sleep quality.

SECONDARY OUTCOMES:
sleep quality | the second postoperative night, third postoperative night
  Richards-Campbell sleep questionnaire (RCSQ) score is used to assess the sleep quality, the total score is 100 point, the lowest score is 0 point, and the highest score is 100 point, with higher scores representing better sleep quality.
Incidence of delirium | from the first to the fifth postoperative day
  Incidence of delirium
pain score(FPS-R) | from the first day to the fifth postoperative day
  Wong-Baker facial expression pain scale revision (FPS-R) at rest and during activity, the lowest score is 0 point, and the highest score is 10 points, with higher scores indicating more severe pain.
pain (NRS) | from the first day to the fifth postoperative day
  Numeric Rating Scale (NRS) at rest and during activity, the total score is 10 points, the lowest score is 0 point, and the highest score is 10 points, with higher scores indicating more severe pain.
drugs | from the first day to the fifth postoperative day
  Additional consumption of analgesic drugs
complications | perioperatively
  Postoperative complications during hospitalization: pulmonary infection, myocardial infarction, renal failure, gastrointestinal bleeding, hypotension, bradycardia, dizziness, nausea, vomiting, nightmares and other psychiatric symptoms
Cognitive function | one month after surgery
  Cognitive function ： Montreal Cognitive Assessment (t-MoCA) score of the telephone version, the total score is 22 points, with a minimum of 0 point and a maximum of 22 points, with higher scores, the cognitive function is better.
Mortality rate | one month after surgery
  Mortality rate
outcomes | one month after surgery
  complications

CONTACTS AND LOCATIONS:
Overall Officials: Tao Luo, MD,PhD, Principal Investigator — Peking University Shenzhen Hospitai
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butris N, Tang E, Pivetta B, He D, Saripella A, Yan E, Englesakis M, Boulos MI, Nagappa M, Chung F. The prevalence and risk factors of sleep disturbances in surgical patients: A systematic review and meta-analysis. Sleep Med Rev. 2023 Jun;69:101786. doi: 10.1016/j.smrv.2023.101786. Epub 2023 Apr 19. PMID 37121133
- [Background] Qiu D, Wang XM, Yang JJ, Chen S, Yue CB, Hashimoto K, Yang JJ. Effect of Intraoperative Esketamine Infusion on Postoperative Sleep Disturbance After Gynecological Laparoscopy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244514. doi: 10.1001/jamanetworkopen.2022.44514. PMID 36454569
- [Background] Su X, Wang DX. Improve postoperative sleep: what can we do? Curr Opin Anaesthesiol. 2018 Feb;31(1):83-88. doi: 10.1097/ACO.0000000000000538. PMID 29120927
- [Background] Myoji Y, Fujita K, Mawatari M, Tabuchi Y. Changes in sleep-wake rhythms, subjective sleep quality and pain among patients undergoing total hip arthroplasty. Int J Nurs Pract. 2015 Dec;21(6):764-70. doi: 10.1111/ijn.12345. Epub 2014 Apr 30. PMID 24779591
- [Background] Driesman AS, Montgomery WC, Kleeman-Forsthuber LT, Johnson RM, Dennis DA, Jennings JM. Perioperative Sleep Quality Disturbances in Total Joint Arthroplasty is Multifactorial. J Arthroplasty. 2024 Jun;39(6):1474-1479. doi: 10.1016/j.arth.2023.12.009. Epub 2023 Dec 8. PMID 38072098
- [Background] Chen H, Fang Z, Wu YY, Zhao CH, Wang YJ, Zhu XH, Cheng XQ. Association between perioperative self-reported sleep disturbances and delirium risk in elderly patients following total joint arthroplasty: a cohort study. J Sleep Res. 2024 Oct;33(5):e14168. doi: 10.1111/jsr.14168. Epub 2024 Feb 21. PMID 38380761
- [Background] Pettit RJ, Gregory B, Stahl S, Buller LT, Deans C. Total Joint Arthroplasty and Sleep: The State of the Evidence. Arthroplast Today. 2024 Apr 24;27:101383. doi: 10.1016/j.artd.2024.101383. eCollection 2024 Jun. PMID 39071825
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Song B, Zhu J. A Novel Application of Ketamine for Improving Perioperative Sleep Disturbances. Nat Sci Sleep. 2021 Dec 25;13:2251-2266. doi: 10.2147/NSS.S341161. eCollection 2021. PMID 34992482
- [Background] Horacek J, Janda R, Gornerova N, Jajcay L, Andrashko V. Several reasons why ketamine as a neuroplastic agent may have failed to prevent postoperative delirium: Implications for future protocols. Neurosci Lett. 2023 Feb 28;798:137095. doi: 10.1016/j.neulet.2023.137095. Epub 2023 Jan 21. PMID 36693556
- [Background] Soffin EM, Gibbons MM, Wick EC, Kates SL, Cannesson M, Scott MJ, Grant MC, Ko SS, Wu CL. Evidence Review Conducted for the Agency for Healthcare Research and Quality Safety Program for Improving Surgical Care and Recovery: Focus on Anesthesiology for Hip Fracture Surgery. Anesth Analg. 2019 Jun;128(6):1107-1117. doi: 10.1213/ANE.0000000000003925. PMID 31094775
- [Background] Zhu Y, Feng W, Kong Q, Sheng F, Li Z, Xu W, Li Q, Han Y, Wu X, Jia C, Guo J, Zhao Y. Evaluating the effects of S-ketamine on postoperative delirium in elderly patients following total hip or knee arthroplasty under intraspinal anesthesia: a single-center randomized, double-blind, placebo-controlled, pragmatic study protocol. Front Aging Neurosci. 2023 Nov 30;15:1298661. doi: 10.3389/fnagi.2023.1298661. eCollection 2023. PMID 38099265
- [Result] Krenk L, Jennum P, Kehlet H. Sleep disturbances after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Nov;109(5):769-75. doi: 10.1093/bja/aes252. Epub 2012 Jul 24. PMID 22831887
- [Result] Shakya H, Wang D, Zhou K, Luo ZY, Dahal S, Zhou ZK. Prospective randomized controlled study on improving sleep quality and impact of zolpidem after total hip arthroplasty. J Orthop Surg Res. 2019 Sep 3;14(1):289. doi: 10.1186/s13018-019-1327-2. PMID 31481074
- [Result] Liu X, Hu X, Li R, Zhang Y. Combination of post-fascia iliaca compartment block and dexmedetomidine in pain and inflammation control after total hip arthroplasty for elder patients: a randomized control study. J Orthop Surg Res. 2020 Feb 10;15(1):42. doi: 10.1186/s13018-020-1562-6. PMID 32041613
- [Result] Shafiei SH, Siavashi B, Ghasemi M, Golbakhsh MR, Baghdadi S. Single High-Dose Systemic Methylprednisolone Administered Preoperatively Improves Pain Control and Sleep Quality After Total Hip Arthroplasty: A Double-Blind, Randomized Controlled Trial. Arthroplast Today. 2022 May 30;16:78-82. doi: 10.1016/j.artd.2022.03.006. eCollection 2022 Aug. PMID 35662994
- [Result] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Result] Chen Z, Tang R, Zhang R, Jiang Y, Liu Y. Effects of dexmedetomidine administered for postoperative analgesia on sleep quality in patients undergoing abdominal hysterectomy. J Clin Anesth. 2017 Feb;36:118-122. doi: 10.1016/j.jclinane.2016.10.022. Epub 2016 Dec 1. PMID 28183547
- [Result] Liu H, Wei H, Qian S, Liu J, Xu W, Luo X, Fang J, Liu Q, Cai F. Effects of dexmedetomidine on postoperative sleep quality: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2023 Mar 21;23(1):88. doi: 10.1186/s12871-023-02048-6. PMID 36944937
- [Result] Zhu S, Liu Y, Wang X, Wang L, Li J, Xue X, Li Z, Liu J, Liu X, Zhao S. Different Sedation Strategies in Older Patients Receiving Spinal Anesthesia for Hip Surgery on Postoperative Delirium: A Randomized Clinical Trial. Drug Des Devel Ther. 2023 Dec 29;17:3845-3854. doi: 10.2147/DDDT.S439543. eCollection 2023. PMID 38169975
- [Result] Ye Q, Hu Y, Xing Q, Wu Y, Zhang Y. The Effects of Opioid-Free Anesthesia with Dexmedetomidine and Esketamine on Postoperative Anesthetic-Related Complications for Hip Surgery in the Elderly. Int J Gen Med. 2024 Dec 17;17:6291-6302. doi: 10.2147/IJGM.S492771. eCollection 2024. PMID 39712198
- [Result] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963
- [Result] Yang JR, Li YY, Ran TJ, Lin XY, Xu JY, Zhou SL, Huang PJ. Esketamine Combined with Dexmedetomidine to reduce Visceral Pain During elective Cesarean Section Under Combined Spinal-Epidural Anesthesia: A double-Blind Randomized Controlled Study. Drug Des Devel Ther. 2024 Jun 18;18:2381-2392. doi: 10.2147/DDDT.S460924. eCollection 2024. PMID 38911034
- [Result] Griffiths R, Babu S, Dixon P, Freeman N, Hurford D, Kelleher E, Moppett I, Ray D, Sahota O, Shields M, White S. Guideline for the management of hip fractures 2020: Guideline by the Association of Anaesthetists. Anaesthesia. 2021 Feb;76(2):225-237. doi: 10.1111/anae.15291. Epub 2020 Dec 2. PMID 33289066
- [Result] Song Y, Liu Y, Yuan Y, Jia X, Zhang W, Wang G, Jia Y, Wang X, Liu L, Li W, Li X, Cai N, Liu C, Li Y, Han Y, Zhou Y, Mi X, Shi C, Wang JQ, Vuylsteke A, Guo X, Li Z. Effects of general versus subarachnoid anaesthesia on circadian melatonin rhythm and postoperative delirium in elderly patients undergoing hip fracture surgery: A prospective cohort clinical trial. EBioMedicine. 2021 Aug;70:103490. doi: 10.1016/j.ebiom.2021.103490. Epub 2021 Jul 17. PMID 34280784